CLINICAL TRIAL: NCT01775046
Title: Post-market Study on Valiant Thoracic Stent Graft With the Captivia Delivery System in the Treatment of Descending Thoracic Aortic Diseases
Brief Title: Valiant Thoracic Stent Graft With the Captivia Delivery System in the Treatment of Descending Thoracic Aortic Diseases (VALIANT CAPTIVIA France)
Status: Completed | Type: Observational
Sponsor: Medtronic Cardiovascular (Industry)
Responsible Party: Sponsor
Other Study IDs: MDTVCFRANCE001
Record Dates: First submitted 2013-01-21; First posted 2013-01-24 (Estimated); Last update posted 2022-02-09 (Actual); Status verified 2022-01

CONDITIONS: Aortic Aneurysm, Thoracic; Descending Thoracic Aortic Dissection; Penetrating Ulcer; Aorta Thoracic; Traumatic Rupture; Aortic Diseases
Keywords: Valiant; Captivia; Stent Graft; Thoracic; Aortic
MeSH Terms: conditions — Aortic Aneurysm, Thoracic; Dissection, Thoracic Aorta; Penetrating Atherosclerotic Ulcer; Aortic Diseases | interventions — Endovascular Aneurysm Repair

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- DTA patients: 160 patients presenting with a disease of descending thoracic aorta(DTA)with an indication for endovascular treatment with Valiant Thoracic Stent Graft with the Captivia Delivery System and who meet the inclusion/exclusion criteria are intended to participate in this non-interventional.
  Interventions: Device: DTA patients (Valiant)

INTERVENTIONS:
Device: DTA patients (Valiant) — Valiant Thoracic Stent Graft Implantation
  Other Names: TEVAR

SUMMARY:
The objective of this study is to assess the benefits of endovascular technique in terms of efficacy and safety of Valiant Thoracic Stent Graft with the Captivia Delivery System in the treatment of thoracic aortic disease, in a cohort of patients representative of the population treated under real-life conditions of use in France for up to 5 years.

DETAILED DESCRIPTION:
Data regarding the use under routine practice of thoracic aortic stent grafts in France are expected by the French National Authority for Health (HAS). Therefore, in its opinion report from December 22, 2009, HAS makes the maintenance of reimbursement approval of each stent graft dependent on the presentation of results of a specific follow-up study carried out in a cohort of patients representative of the French population treated under real-life conditions of use. This prospective cohort study must involve patients implanted after registration on the LPPR (List of Products and Services qualifying for Reimbursement). The results of the follow-up study must be forwarded to the National Committee for Evaluation of Medical Devices and Health Technologies (CNEDiMTS) for examination once a year. The assessment of this follow-up could lead to the recommendation by CNEDiMTS to continue or stop the reimbursement of the concerned stent graft.

In France, The Valiant Thoracic Stent Graft with the Captivia Delivery System is registered on the LPPR for a period of 3 years since January 12, 2011. In order to comply with HAS expectations, Medtronic Bakken Research Center is setting up this long term non-interventional study on the Valiant Thoracic Stent Graft with the Captivia Delivery System.

ELIGIBILITY:
Inclusion Criteria:

* Any patient requiring placement of the Valiant Thoracic Stent Graft for the treatment of a disease of his/her descending thoracic aorta.
* Patient or holder of parental authority not opposed to the collection and release of the personal information required by the study.
* Patient or holder of parental authority has consented for study participation and the Medtronic approved Data Release Form has been signed and personally dated by patient or holder of parental authority and by the investigator.

Exclusion Criteria:

* Patient in whom clinical follow-up will not be possible i.e. patient not able to come back for follow-up visits (ex. patient living abroad).
* Prior implantation of a thoracic stent graft.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Subjects diagnosed with a disease of descending thoracic aorta (DTA) and requiring endovascular treatment with Stent Graft.
Sampling Method: Non-Probability Sample
Enrollment: 160 (Actual)
Dates: Start 2013-03-23 (Actual); Primary Completion 2021-06-21 (Actual); Study Completion 2021-12-09 (Actual)

PRIMARY OUTCOMES:
All-cause mortality | 5 years

SECONDARY OUTCOMES:
Exclusion of aneurysm, penetrating aortic ulcer (PAU), false lumen or rupture site | Through 5 years
Major Adverse Events | Through 5 years
  This includes respiratory, neurological, vascular, cardiac, renal, bleeding, visceral and infectious complications and any complication leading to death
Conversion to open repair | Through 5 years
Endovascular or surgical secondary procedures | Through 5 years
Adverse device effects | Through 5 years
Thoracic disease-related mortality | Through 5 years

CONTACTS AND LOCATIONS:
Overall Officials: Hervé Rousseau, MD, PhD, Principal Investigator — CHU Rangueil, 1 Avenue Jean Poulhes, TSA 50 032, 31059 TOULOUSE Cedex 9, FRANCE
Locations (17):
- France (17):
  - CHU Amiens Picardie, Hôpital Sud, Amiens
  - CHU de Bordeaux, Groupe Hospitalier Pellegrin, Bordeaux
  - Hôpital Henri Mondor, Créteil
  - CHU Grenoble, Hôpital A. Michallon, La Tronche
  - Hôpital Privé de Parly 2, Le Chesnay
  - Centre Chirurgical Marie Lannelongue, Le Plessis-Robinson
  - CHU de Limoges, Limoges
  - Hôpital Privé Vert Coteau, Marseille
  - Hôpital de la Timone, Marseille
  - Hôpital Nord, Marseille
  - Hôpital Européen Georges Pompidou, Paris
  - Hôpital Pitié Salpêtrière, Paris
  - Clinique Belledonne, Saint-Martin-d'Hères
  - CHU de Saint-Etienne, Hôpital Nord, Saint-Priest-en-Jarez
  - CHU Rangueil, Toulouse
  - Clinique Pasteur, Toulouse
  - Clinique du Tonkin, Villeurbanne

IPD SHARING:
Plan to Share IPD: No
Only multi center data will be available